CLINICAL TRIAL: NCT01645397
Title: Exhaled Nitric Oxide and Airway Caliber in Children With Asthma
Status: Completed | Type: Observational
Sponsor: Atlantic Health System (Other)
Responsible Party: Principal Investigator, Patricia Breitwieser, Coordiantor, Respiratory Center for Children, Atlantic Health System
Other Study IDs: R10-06-013
Record Dates: First submitted 2011-06-23; First posted 2012-07-20 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2014-01

CONDITIONS: Asthma in Children
Keywords: Asthma; Deep inhalation; Exhaled nitric oxide
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Asthma, elevated exhaled NO: Children with asthma with elevated exhaled NO at initial evaluation (>25ppb)

SUMMARY:
The purpose of this study is to assess if in steroid naïve asthmatic children with elevated baseline exhaled nitric oxide, treatment with inhaled steroid and normalization of exhaled nitric oxide level results in restoration of the bronchodilator response to deep inhalation.

DETAILED DESCRIPTION:
Previous studies have shown that a deep inhalation (DI) would increase airway caliber in normal subjects. Whereas in asthmatics with spontaneous bronchoconstriction (obstruction of the airway), DI was shown to worsen airway obstruction. The mechanism for this variability in response to DI is not well-understood, but seems to be a key in understanding the pathophysiology of the disease, and possibly in the development of an effective therapy. Air way inflammation resulting in airway wall thickening and peribronchial edema is thought to play a role how the airway responds to deep inhalation. This study assess if reduction in airway inflammation (as measured by level of exhaled NO)results in optimization of the bronchodilator response to deep inhalation

ELIGIBILITY:
Inclusion Criteria:

* Age: > 6 years at age of screening.
* Physician diagnosed asthma
* Elevated exhaled NO at initial evaluation (>25ppb)
* Be able to reproducibly perform DI maneuvers and all other pulmonary function testing
* Be clinically stable for at least 2 weeks prior to screening with no evidence of acute upper or lower respiratory infection or current pulmonary exacerbation.
* Has not been on inhaled or oral steroid for at least 4 weeks prior to enrollment in the study.
* Parent/child willingness to enroll in the study and provide written informed consent.
* Be able to present for the required study visits.

Exclusion Criteria:

* Chest wall or spinal column deformity; known cardiac, neuromuscular, or other chronic diseases
* Use of beta agonist, theophylline, leukotriene receptor antagonists, or caffeine-containing soft drinks 12 hr prior to the study.
* Use of inhaled steroid in the past 4 weeks.
* Respiratory infection or asthma exacerbation in the previous 2 weeks

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children, six years of age or older, with asthma attending asthma clinic
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-06; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change in M/P40 ratio from baseline at 4 weeks of treatment with inhaled steroid | at baseline and 4 weeks later
  M/P40 ratio is defined as the ratio of flow at 40% of FVC (forced vital capacity) on the flow-volume curve after maximal inspiration to flow at 40% of FVC on the flow-volume curve after partial (60%-70% of FVC) inspiration (M/P40 ratio)

SECONDARY OUTCOMES:
Change in Ratio of post DI to pre DI airway resistance from baseline at 4 weeks of treatment with inhaled steroid | at baseline and 4 weeks later
  Post-DI to pre-DI airway resistance at 5 Hz (R5) ratio (as measured by impulse oscillometry) from baseline (elevated exhaled NO) to 4-6 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Dagnachew Assefa, MD, Principal Investigator — Atlantic Health System
Locations (1):
- Goryeb Children's Hospital, Atlantic Health, Morristown, New Jersey, United States